CLINICAL TRIAL: NCT04480203
Title: Coping After Breast Cancer - CABC - Stressmestring Etter Brystkreft - SEB
Brief Title: Coping After Breast Cancer - a Randomized Clinical Trial With Two Digital Interventions
Acronym: CABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CABC - Kreftfor project - SEB
Record Dates: First submitted 2020-07-09; First posted 2020-07-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer Patients; Health, Subjective
Keywords: Health Related Quality of Life; Stress management intervention

STUDY DESIGN:
Intervention Model Description: An intervention study of breast cancer patients with two digital intervention arms and one control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the staff that have contact with the participants will know who receives which intervention. The statistician and investigators will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive based stress management (CBSM) (Active Comparator): Cognitive based digital intervention.
  Interventions: Other: Stressproffen cognitive based stress management
- Mindfulness based intervention (MBI) (Active Comparator): Mindfulness based digital intervention.
  Interventions: Other: Stressproffen mindfulness based intervention
- Control (Placebo Comparator): Control arm. No intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Stressproffen cognitive based stress management — The participants will download an app (Stressproffen 2A) with cognitive based stress management.
  Other Names: CBSM
  Arms: Cognitive based stress management (CBSM)
Other: Stressproffen mindfulness based intervention — The participants will download an app (Stressproffen 2B) with mindfulness based intervention.
  Other Names: MBI
  Arms: Mindfulness based intervention (MBI)
Other: Control — The participants will receive no app. (They will be able to download it after the end of the 3 year study).
  Arms: Control

SUMMARY:
1. Breast cancer patients and age-matched controls are first invited to answer questions on HRQoL.
2. Among responding breast cancer patients, a subset are invited in a randomized clinical trial with two digital interventions for cancer stress management, cognitive based stress management (CBSM) and mindfulness based intervention (MBI), as well as a control group.
3. The goal is to determine whether digital CBSM or MBI can effectively reduce stress levels as compared to a control group. Second, whether these interventions can improve HRQoL (or avoid onset of HRQoL problems) for patients with breast cancer, compared to a control group.

DETAILED DESCRIPTION:
After completing the baseline HRQoL assessment, eligible breast cancer patients will be invited to participate in a randomized clinical trial.

Those who are willing will be randomly allocated to one of the following arms: a) Digital cognitive based stress management, b) Digital mindfulness based intervention or c) Control group.

The intervention is based on a revised version of the Stressproffen app, which was developed by the Oslo University Hospital (Lise Solberg Nes, Elin Børøsund and others).

Outcome measures include measures of perceived stress and HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* first occurrence breast cancer diagnosed from Jan 1, 2020
* non-metastatic cancer stage 0-III

Invasive tumors must be:

* HER2 positive (regardless of ER, PR) or
* ER negative
* (may later include other ER+ if not conflict with recruitment for EMIT/OPTIMA)

Exclusion Criteria:

* None

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 390 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress | change from CABC baseline (week 0) to f-up week 21
  Cohens perceived stress scale. Unit is summary score.

SECONDARY OUTCOMES:
Subjective health (HRQoL) | change from CABC baseline (week 0) to f-up week 21
  RAND-36 questionnaire. Unit is summary score and module-specific scores
Coping | change from CABC baseline (week 0) to f-up week 21
  TOMCATS questionnaire. Unit is summary score.
Anxiety and depression | change from CABC baseline (week 0) to f-up week 21
  PHQ-4 questionnaire. Unit is summary score.
Fatigue | change from CABC baseline (week 0) to f-up week 21
  Chalders' fatigue questionnaire. Unit is summary score.
Mindfulness | change from CABC baseline (week 0) to f-up week 21
  Baer 2006 mindfulness questionnaire. Unit is summary score.
Sleep | change from CABC baseline (week 0) to f-up week 21
  selected questions fro SUSSH questionnaire. Unit is summary score.
EORTC QLQ-C30 | From NBCR baseline to f-up week 20
  EORTC health related quality of life (HRQoL) general questionnaire. Unit is summary score.
EORTC QLQ-BR23 | From NBCR baseline to f-up week 20
  EORTC breast cancer questionnaire. Unit is summary score.
Neuropathy (FACT GOG-NTX and -ES) | From NBCR baseline to f-up week 20
  neuropathy questionnaire. Unit is summary score.
Stress | change from CABC baseline (week 0) to f-up month 15
  Cohens perceived stress scale. Unit is summary score.
Subjective health (HRQoL) | change from CABC baseline (week 0) to f-up month 15
  RAND-36 questionnaire. Unit is summary score and module-specific scores
Coping | change from CABC baseline (week 0) to f-up month 15
  TOMCATS questionnaire. Unit is summary score.
Fatigue | change from CABC baseline (week 0) to f-up month 15
  Chalders' fatigue questionnaire. Unit is summary score.
Mindfulness | change from CABC baseline (week 0) to f-up month 15
  Baer 2006 mindfulness questionnaire. Unit is summary score.
Anxiety and depression | change from CABC baseline (week 0) to f-up month 15
  PHQ-4 questionnaire. Unit is summary score.
Sleep | change from CABC baseline (week 0) to f-up month 15
  selected questions fro SUSSH questionnaire. Unit is summary score.
Work | status at f-up month 15
  questions on employment. Whether employed and percentage
Stress | change from CABC baseline (week 0) to f-up month 27
  Cohens perceived stress scale. Unit is summary score.
Subjective health (HRQoL) | change from CABC baseline (week 0) to f-up month 27
  RAND-36 questionnaire. Unit is summary score and module-specific scores
Coping | change from CABC baseline (week 0) to f-up month 27
  TOMCATS questionnaire. Unit is summary score.
Anxiety and depression | change from CABC baseline (week 0) to f-up month 27
  PHQ-4 questionnaire. Unit is summary score.
Fatigue | change from CABC baseline (week 0) to f-up month 27
  Chalders' fatigue questionnaire. Unit is summary score.
Mindfulness | change from CABC baseline (week 0) to f-up month 27
  Baer 2006 mindfulness questionnaire. Unit is summary score.
Sleep | change from CABC baseline (week 0) to f-up month 27
  selected questions fro SUSSH questionnaire. Unit is summary score.
EORTC QLQ-C30 | change from NBCR baseline to f-up month 27
  EORTC health related quality of life (HRQoL) general questionnaire. Unit is summary score.
EORTC QLQ-BR23 | change from NBCR baseline to f-up month 27
  EORTC breast cancer questionnaire. Unit is summary score.
Neuropathy (FACT GOG-NTX and -ES) | From NBCR baseline to f-up month 27
  neuropathy questionnaire. Unit is summary score.

CONTACTS AND LOCATIONS:
Overall Officials: Giske Ursin, MD, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svendsen K, Nes LS, Leithe S, Meland A, Gjelsvik YM, Borosund E, Larsson IM, Myklebust TA, Balto A, Rygg CM, Kiserud CE, Antoni MH, Chalder T, Mjaaland I, Carlson LE, Eriksen HR, Ursin G. Testing two digital stress-management interventions in a randomized controlled trial of breast cancer patients. Sci Rep. 2025 Nov 6;15(1):38966. doi: 10.1038/s41598-025-22889-0. PMID 41198868
- [Derived] Svendsen K, Nes LS, Meland A, Larsson IM, Gjelsvik YM, Borosund E, Rygg CM, Myklebust TA, Reinertsen KV, Kiserud CE, Skjerven H, Antoni MH, Chalder T, Mjaaland I, Carlson LE, Eriksen HR, Ursin G. Coping After Breast Cancer: Protocol for a Randomized Controlled Trial of Stress Management eHealth Interventions. JMIR Res Protoc. 2023 May 24;12:e47195. doi: 10.2196/47195. PMID 37103493